CLINICAL TRIAL: NCT01623271
Title: Treatment of Complex Regional Pain Syndrome With Once Daily Gastric-Retentive Gabapentin (Gralise)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to limited population of research participants.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jianren Mao, MD, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012P000466
Record Dates: First submitted 2012-06-12; First posted 2012-06-19 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Complex Regional Pain Syndrome I (CRPS I)
Keywords: CRPS I
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CRPS I Pain Subjects (Experimental): This is an open label study that involves taking Gralise pills (gastic-retentive gabapentin) for 8 weeks.
  Day 1-15: Titration phase- titrate Gralise from 300 mg/day to 1800 mg/day Day 16-42: Maintenance phase- maintain the dose of 1800 mg/day Day 43-56: Taper phase- taper the Gralise from 100 mg/day to 300 mg/day
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin
  Other Names: Gralise

SUMMARY:
The purpose of this study is to see if an FDA-approved drug (Gralise) can help people with certain types of neuropathic pain without causing too many side effects.

DETAILED DESCRIPTION:
This research is being conducted to see if the drug Gralise can help people with Complex Regional Pain Syndrom Type I (CRPS I) without causing too many side effects. CRPS I is one of the most common conditions of neuropathic pain (pain that results from damage to nerves in the peripheral nervous system). Gralise is approved by the U.S. Food and Drug Administration (FDA) to treat postherpetic neuralgia (a complication of the disease Shingles, which is caused by the chickenpox virus), but is not approved to treat CRPS I.

ELIGIBILITY:
Inclusion Criteria:

1. Subject will be between 18 to 80 years of age.
2. Subject has not been on Gralise.
3. Subject has not been on gabapentin for at least one month.
4. Subject agrees to make no change in his/her current pain medications during the study period to ensure that comparisons can be made before and after the Gralise treatment.
5. Subject has a VAS pain score of 5 or above at the beginning of the study.
6. Subject has had CRPS I for at least three months to avoid clinical uncertainty and minimize the study variation.
7. Female subjects of childbearing age must have a negative urine pregnancy test at the initial visit.

Exclusion Criteria:

1. Subject has severe liver or renal disease that will affect the elimination of Gralise. (Renal dysfunction is defined as eGFR < 60. Hepatic dysfunction is defined as LFTs ≥ 3X ULN.)
2. Subject has pending litigation related to his/her CRPS I condition.
3. Subject is pregnant or lactating.
4. Subject is allergic to gabapentin or Gralise.
5. Subject has a positive urine (illicit) drug test.
6. Subject has any history of suicidal thoughts or behaviors, as self reported or in documented medical history.
7. Subjects with known seizure disorders (except febrile seizures) and/or taking antiepileptic drugs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jianren Mao, M.D., Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mao J. Translational pain research: achievements and challenges. J Pain. 2009 Oct;10(10):1001-11. doi: 10.1016/j.jpain.2009.06.002. Epub 2009 Jul 22. PMID 19628433
- [Result] Mao J, Chen LL. Systemic lidocaine for neuropathic pain relief. Pain. 2000 Jul;87(1):7-17. doi: 10.1016/S0304-3959(00)00229-3. PMID 10863041
- [Result] Mao J, Gold MS, Backonja MM. Combination drug therapy for chronic pain: a call for more clinical studies. J Pain. 2011 Feb;12(2):157-66. doi: 10.1016/j.jpain.2010.07.006. Epub 2010 Sep 17. PMID 20851058
- [Result] Sindrup SH, Jensen TS. Efficacy of pharmacological treatments of neuropathic pain: an update and effect related to mechanism of drug action. Pain. 1999 Dec;83(3):389-400. doi: 10.1016/S0304-3959(99)00154-2. PMID 10568846
- [Result] van de Vusse AC, Stomp-van den Berg SG, Kessels AH, Weber WE. Randomised controlled trial of gabapentin in Complex Regional Pain Syndrome type 1 [ISRCTN84121379]. BMC Neurol. 2004 Sep 29;4:13. doi: 10.1186/1471-2377-4-13. PMID 15453912

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CRPS I Pain Subjects
Started | 5
Completed | 3
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | CRPS I Pain Subjects
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Visual Analog Scale (VAS) [Mean (Full Range); unit: units on a scale] — Pain score on a scale of 0-10
  units on a scale | 5.8 [3 to 9]

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) at Visit 3
Description: Subjects rated their pain using the VAS at visit 3, which was the last day of their maintenance phase. After this visit, subjects begin to taper the gralise. The VAS is subject reported on a scale of 0-10 with 0 being no pain and 10 being the worst pain they can imagine. Results reported are an average of the 3 subjects who completed visit 3.
Time Frame: At visit 3
Population: Only 3 subjects completed visit 3. The other 2 subjects dropped out due to expected side effects.
Measure: Mean (Standard Deviation); unit: units on the VAS
Arm/Group | CRPS I Pain Subjects
Number analyzed (Participants) | 3
units on the VAS | 3.67 (1.15)
Statistical Analysis 1: Comparison: CRPS I Pain Subjects; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | CRPS I Pain Subjects
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRPS I Pain Subjects (N=5)
Expected Side Effects of Gralise (General disorders) | 2 (2) — - Headache, nausea, dizziness, fatigue, increased joint pain

LIMITATIONS AND CAVEATS:
Problems with recruitment and early termination of the study consequently resulted in uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes